CLINICAL TRIAL: NCT04608058
Title: Comparison of Self-management Behaviors Education Through Digital Storytelling Method and Conventional Method in Adolescents With Type 1 Diabetes Referred to Diabetes Clinic in Hospitals Affiliated to Shiraz University of Medical Sciences.
Brief Title: Promoting Self-management Behaviors in Adolescents With Type 1 Diabetes, Using Digital Storytelling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nahid Zarifsanaiey (Other)
Responsible Party: Sponsor-Investigator, Nahid Zarifsanaiey, Associate Professor, Shiraz University of Medical Sciences
Organization: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1398.244
Record Dates: First submitted 2020-10-27; First posted 2020-10-29 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 1; Self-Management
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): At first, participants' demographic data, the levels of "self-management", and "HbA1c "were documented at the commencement of the study. Then, asynchronous Diabetes self-management training, using digital storytelling was made available to this group. Post-test data were collected 3 months after the pretest.
  Interventions: Behavioral: Digital storytelling training
- No Intervention (Experimental): At first, participants' demographic data, the levels of "self-management", and "HbA1c "were documented at the commencement of the study. Then, the control group received the clinics' routine training. Post-test data were collected 3 months after the pretest.
  Interventions: Behavioral: Routine training

INTERVENTIONS:
Behavioral: Digital storytelling training — The digital content in this study is called "Diabetes and Bumblebee". It features 35 minutes of animation that provides children with a brief description of the disease, its symptoms and complications, treatment methods, the type of insulin, how to preserve insulin, the importance of nutrition and exercise in treating diabetes as well as efficient communication and collaboration with parents and healthcare providers. Exciting and interactive animations were used to depict the daily life of a adolescence with diabetes.
  Arms: Intervention
Behavioral: Routine training — The control group received the clinics' routine training include face to face class education.
  Arms: No Intervention

SUMMARY:
The aim of this study was to evaluate the effects of digital storytelling on the Self-Management behavior of adolescents with type 1 diabetes (TID).

DETAILED DESCRIPTION:
In this single-blind randomized controlled trial, 60 eligible adolescents with TID were selected based on a convenient sampling method. Next, the participants were randomly allocated into two parallel groups: intervention (training with digital storytelling method, n=30) or control (training with conventional) n=30) groups. Before and three months after the intervention the patients' levels of self-management behaviors according to Self-Management of TID amongst adolescents (SMOD-A); in addition to the Glycated Hemoglobin test (HbA1c) were measured.

ELIGIBILITY:
Inclusion Criteria:

* adolescents with TID
* using medication (insulin)
* willing to participate in the study and complete the informed consent
* having a basic knowledge of working with computers
* ability to communicate on the telephone.

Exclusion Criteria:

* physical or mental disabilities
* take anti-anxiety or antidepressant medication

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Self-management behavior | 3 months
  Self-Management of TID in Adolescence (SMOD-A) questionnaire which includes 48 items in 5 domains; cooperation with Parents, Diabetes care activities, Diabetes Problem-Solving, Diabetes Communication, and Goal in Diabetes. Each item is scored on a 4-point Likert scale ranging from 0 (never) to 3 (always). Higher scores are associated with better self-management behaviors.

SECONDARY OUTCOMES:
Change in Glycated hemoglobin A1c | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nahid zarifsanaiey, Principal Investigator — associate Professor, Virtual school, Shiraz University of Medical Sciences, Shiraz, Iran.
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: Undecided